CLINICAL TRIAL: NCT05045378
Title: Low-dose Ketamine Infusion Among Adolescents With Treatment-resistant Depression: a Randomized, Double-blind Placebo-control Study
Brief Title: Low-dose Ketamine Infusion Among Adolescents With Treatment-resistant Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-02-015A
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2022-04

CONDITIONS: Treatment-resistant Depression; Major Depressive Disorder
Keywords: adolescent; ketamine; N-methyl-D-aspartate receptor (NMDAR) antagonist
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major | interventions — Midazolam; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. Two 0.045mg/kg midazolam infusions (Active Comparator): Two 0.045mg/kg midazolam infusions as active placebo
  Interventions: Drug: Midazolam (active placebo)
- 2. First 0.045mg/kg midazolam infusion and Second 0.5mg/kg ketamine infusion (Experimental): Single ketamine infusion + Single midazolam placebo infusion
  Interventions: Drug: Ketamine and Midazolam (active placebo)
- 3. Two 0.5mg/kg ketamine infusions (Experimental): Repeated (Two) ketamine infusions: Two 0.5mg/kg ketamine infusions
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Midazolam (active placebo) — Arm1: Two 0.045mg/kg midazolam infusions at Day1 and Day3。
  Arms: 1. Two 0.045mg/kg midazolam infusions
Drug: Ketamine and Midazolam (active placebo) — Arm2: First 0.045mg/kg midazolam infusion and Second 0.5mg/kg ketamine infusion。
  Arms: 2. First 0.045mg/kg midazolam infusion and Second 0.5mg/kg ketamine infusion
Drug: Ketamine — Arm3: Two 0.5mg/kg ketamine infusions。
  Arms: 3. Two 0.5mg/kg ketamine infusions

SUMMARY:
In the past decades, the prevalence of adolescent depression and suicide increased significantly in Taiwan and worldwide. To date, the suicide mortality is the second mortality cause in the adolescent and young adult population in Taiwan. Previous studies reported that up to 40% of adolescents with major depressive disorder did not respond to at least two traditional antidepressants with the optimal dose and adequate duration. Those patients would be considered the cases with treatment-resistant depression (TRD), which is related to the poor prognosis, chronic depressive course, higher suicidal risk, severer cognitive dysfunction, and greater family burdens. However, much less studies investigated the treatment strategy for adolescent TRD compared with that for adult TRD. In this decade, low-dose ketamine infusion has been proved as a rapid-acting antidepressant for adult patients with TRD. In recent 5 years, the investigators study team finished two randomized, double-blind, and placebo-control trials to support the rapid antidepressant and anti-suicidal effect in Taiwanese adult patients with TRD. The investigators published several SCI studies about the investigators clinical findings and the underlying brain mechanisms. In the following 4 years, the investigators will conduct a new randomized, double-blind, and placebo-control trial in the adolescent TRD. It will be the first clinical trial for ketamine effect in adolescent TRD worldwide. The investigators will enroll 54 adolescents aged between 13 and 29 with TRD in four years. The investigators hypothesize that low-dose ketamine will be effective and well tolerable for adolescents with TRD.

DETAILED DESCRIPTION:
1. Treatment-resistant depression (TRD) in adolescence:

   Major depressive disorder (MDD) in adolescents is characterized by a high risk of suicidality, recurrence, and chronicity and has been a topic of concern for decades in the fields of public health and clinical psychiatry (Goodyer, Dubicka et al. 2007; Garber and Weersing 2010). The estimated prevalence of MDD is 8%-20% in the adolescent population (Yorbik, Birmaher et al. 2004; Thapar, Collishaw et al. 2012). Longitudinal studies on community-based and clinic-based population samples have suggested that 60%-90% of adolescents reported to have depression achieve remission within a year; moreover, follow-up studies have indicated that 50% to 70% of patients who remit report subsequent depressive episodes within 5 years (Dunn and Goodyer 2006; Thapar, Collishaw et al. 2012).

   Relevant studies have reported that adolescents with depression have less response to antidepressants and lower remission rates than adults with depression, which may indicate a higher prevalence of TRD in adolescent population (Michael and Crowley 2002; Kennard, Silva et al. 2009; Zhou, Michael et al. 2014). The Treatment for Adolescents with Depression Study (TADS) reported that the remission rate following 12-week antidepressant monotherapy or combination treatment using antidepressants and cognitive-behavioral therapy (CBT) was approximately 60% in adolescents with MDD, which may indicate that at least one-third of adolescents with MDD did not respond to treatment or achieve remission after adequate antidepressant, CBT, or combined treatment (Kennard, Silva et al. 2009). The Adolescent Depression, Antidepressants, and Psychotherapy Trial reported that only 57% of adolescents with depression exhibited moderate or substantial improvement after 28 weeks of SSRI or CBT treatment and that up to 20% demonstrated no improvement (Goodyer, Dubicka et al. 2007). Furthermore, Curry et al. evaluated the predictors of response to fluoxetine treatment in adolescents with depression and reported that those with more psychiatric comorbidities, including anxiety disorders, attention deficit hyperactivity disorder (ADHD), and disruptive behavioral disorders, were less likely to benefit from treatment than their counterparts (Curry, Rohde et al. 2006). Hilton et al. further investigated the efficacy of changing antidepressant treatment to another selective serotonin reuptake inhibitor (SSRI) or venlafaxine in adolescents with SSRI-resistant depression and determined that those who did not achieve remission exhibited increased anxiety, ADHD, and behavioral symptoms than those who did (Hilton, Rengasamy et al. 2013).

   However, current guidelines for TRD in adolescent patients with depression remain inadequate despite the high morbidity and severe impairment in these young patients (Zhou, Michael et al. 2014). A recent meta-analysis showed that the overall response rate for the active treatments, including the combination therapy with psychotherapy or second antidepressants, augmentation therapy with lithium/atypical antipsychotics, or the antidepressant-switching, was only 46% among adolescent patients with TRD. Approximately half of the adolescents who presented with TRD responded to active treatment, which suggests that practitioners should remain persistent in managing these challenging cases (Zhou, Michael et al. 2014). Treatment of Resistant Depression in Adolescents (TORDIA) study further suggested that the current clinical guidelines, which recommend pursuing a given treatment strategy for at least 8-12 weeks, may need to be revisited because their data support more vigorous intervention earlier in the course of treatment for nonresponding patients (Emslie, Mayes et al. 2010).
2. Suicide in adolescence:

   The suicide rates in the last half century increased by 60% worldwide, it is estimated that by 2020, suicide would account more than 1 million deaths. The WHO reports that Taiwan is one of the countries with the highest prevalence of suicide mortality (>13/100,000) worldwide (2012; Fazel, Wolf et al. 2013). In Taiwan, the prevalence of suicide mortality reached a peak in 2006 (19.3/100,000). The Taiwan suicidal prevention program was implemented in 2005, and in the following years (2008~2011), the prevalence of suicide mortality declined gradually to 15.1/100,000. But, the prevalence of suicide mortality rebounded up to 16.2/100,000 again in 2012 (Cicinelli, Pasqualetti et al. 2003). More than suicide mortality and committed suicide, the suicide attempt and suicide ideation also gained the clinical and public health attention and concerns in this decades (2012; Fazel, Wolf et al. 2013).

   Suicide among adolescents has gained substantial clinical attention in the psychiatric field in the recent decade and has become a major public health concern worldwide (2012; Fazel, Wolf et al. 2013). The U.S. National Institute of Mental Health reported that suicide was the country's third leading cause of mortality among adolescents and young adults aged 15 to 24 years (2012; Fazel, Wolf et al. 2013). In Taiwan, the Ministry of Health and Welfare indicated that suicide was the second leading cause of mortality among adolescents and young adults, accounting for the death of 7.1/100,000 adolescents and young adults (Cicinelli, Pasqualetti et al. 2003).

   A Taiwan report in 2013, a nationally representative sample of 2835 college students, demonstrated that a surprisingly high prevalence of college students (about 12% of females and 9% of males) had at least one time of attempted suicide in the preceding 12 months (Chou, Ko et al. 2013). Previous studies have demonstrated that more than 70% of adolescents and young adults who attempt suicide or have suicidal ideation have psychiatric disorders, including major depressive disorder, bipolar disorder, anxiety disorders, disruptive behavior disorders, and alcohol and substance use disorders (Brent, Perper et al. 1994; Gould, King et al. 1998; Kelly, Cornelius et al. 2002; Hauser, Galling et al. 2013). Any form of suicide, including suicide ideation, suicide attempt, and suicide mortality, would cause a great amount of physical, mental, and financial loss and burden to the sufferers, the family, the community, and the society. Furthermore, those suicide ideators and suicide attempters remain vulnerable to costly health and social problems in their later life.
3. Low-dose ketamine infusion in adolescent depression:

Based on the higher treatment resistance and the greater suicidal risk in adolescent depression, increasing evidence suggests the potential therapeutic effect of low-dose ketamine infusion in adolescent patients with TRD although there was no any randomized, double-blind, placebo-control clinical trial to investigate this important clinical topic until now. Ketamine is safe, tolerable, and commonly used in the pediatric anesthesia in the past decades (Brewer, Davidson et al. 1972; Raju 1980; Green, Klooster et al. 2001; Koruk, Mizrak et al. 2010). In 2017, Dwyer et al reported the first case report study for the ketamine infusion as a treatment for adolescent depression (Dwyer, Beyer et al. 2017). They described the personal history and clinical course of this case: this patient was considered to be at high risk for suicide. He had a history of three serious suicide attempts involving near-lethal antifreeze ingestion, dextroamphetamine overdose, and self-strangulation. He presented as hopeless about the prospect of psychiatric improvement and complained of persistent thoughts of wanting to die. The patient had failed multiple levels of care (outpatient, intensive outpatient, and residential) and multiple antidepressant medications, with treatment informed by current practice parameters. This patient received intravenous infusions of ketamine, dosed at 0.5 mg/kg over 40 minutes. This patient received 3 infusions during the first week and weekly treatments thereafter, resulting in 7 infusions over an 8-week hospitalization (days 1, 3, 7, 14, 21, 28, 50). At 1 day after his first infusion, he experienced a rapid reduction in his depressive symptoms (61% MADRS reduction; 32% CDRS reduction), suicidal ideation (88% SSI-5 reduction), and hopelessness (57% BHS reduction). The patient had an acute recovery with ketamine treatment, as has been described in adults (Figure 4). He tolerated all infusions well, experiencing mild nausea and mild intrainfusion dissociative symptoms (maximum CADSS of 7 [of a possible 92], which returned to 0 by 80 minutes) (Dwyer, Beyer et al. 2017).

This is a double-blind, randomized-controlled trial of ketamine infusion to test whether 0.5mg/kg ketamine infusion is a safe and effective add-on treatment for adolescents with TRD.

ELIGIBILITY:
Inclusion Criteria:

1. Major depressive episode including unipolar and bipolar depression, according to DSM- 5 criteria and MINI-adolescent version (Mini-International Neuropsychiatric Interview; MINI) diagnostic interview.
2. Age 13 to 19 years old.
3. Body weigh ≧ 30 kg.
4. Treatment-resistant depression, which is defined as poor or unsatisfactory response to at least two different antidepressants administered at an adequate dosage and for an adequate treatment duration
5. Still prominent depressive symptoms with at least 4-week treatment of medication treatment or psychotherapy
6. Voluntary patients and their parents or guardians with signed informed consent proved by institutional review board (IRB)

Exclusion Criteria:

1. Major medical conditions (e.g., head injury, epilepsy, severe renal diseases and cancer).
2. Other axis I psychiatric disorders such as schizophrenia, delusional disorder, organic brain syndrome, and dementia.
3. Pregnancy.
4. Substance abuse in previous 6 months such as cocaine, marijuana, opium, ketamine, PCP (phencyclidine)。
5. Current use of NMDA receptor antagonist (Amantadine, Rimantadine, Lamotrigine, Memantine, Dextromethorphan)
6. Alcohol abuse / dependence within 6 months.
7. Attempt suicide in hospital.
8. Allergy to ketamine
9. Abnormal liver function in recent 3 months。
10. Abnormal ECG (i.e.:arrhythmia)。
11. Fever or infection in recent 5 days。

Ages: 13 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in depressive symptoms measured by Montgomery-Åsberg Depression Rating Scale (MADRS) in adolescents with treatment-resistant depression. | clinical visit or telephone visit evaluation times are Day 1, 2, 3, 4, 5, 6, 7, 14, and 28
  Higher MADRS score indicates more severe depression. The overall score ranges from 0 to 60.
Changes in depressive symptoms measured by Hamilton Rating Scale for Depression (HAMD) in adolescents with treatment-resistant depression. | clinical visit or telephone visit evaluation times are Day 1, 2, 3, 4, 5, 6, 7, 14, and 28
  Higher HAMD score indicates more severe depression. The overall score ranges from 0 to 52.
Changes in depressive symptoms measured by Children's Depression Rating Scale-Revised (CDRS-R) in adolescents with treatment-resistant depression. | clinical visit or telephone visit evaluation times are Day 1, 2, 3, 4, 5, 6, 7, 14, and 28
  Higher CDRS-R score indicates more severe depression. The overall score ranges from 17 to 113.

CONTACTS AND LOCATIONS:
Overall Officials: Mu-Hong Chen, M.D., Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taiwan, Taipei, Taiwan